CLINICAL TRIAL: NCT04122287
Title: Helicobacter Pylori First-line Treatment Containing Tetracycline in Patients Allergic to Penicillin:a Prospective Randomized Controlled Study
Brief Title: Helicobacter Pylori First-line Treatment in Patients Allergic to Penicillin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-SDU-QILU-G709
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Helicobacter Pylori Infection
Keywords: Allergic; Penicillin; Helicobacter pylori; Eradication; Tetracycline
MeSH Terms: interventions — Levofloxacin; Tinidazole

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- levofloxacin-tetracycline-containing quadruple group (Experimental): patients in levofloxacin-tetracycline-containing quadruple group will receive lansoprazole 30mg po bid, tetracycline 500mg po qid , bismuth subcitrate (Colloidal Bismuth Pectin) 200mg po bid, and levofloxacin 500mg po qd for 14d
  Interventions: Drug: Levofloxacin
- tinidazole-tetracycline-containing quadruple group (Active Comparator): patients in tinidazole-tetracycline-containing quadruple group will receive lansoprazole 30mg po bid, tetracycline 500mg po qid , bismuth subcitrate (Colloidal Bismuth Pectin) 200mg po bid, and tinidazole 500mg po tid for 14d.
  Interventions: Drug: tinidazole

INTERVENTIONS:
Drug: Levofloxacin — levofloxacinn-tetracycline-containing quadruple regimens
  Arms: levofloxacin-tetracycline-containing quadruple group
Drug: tinidazole — tinidazole-tetracycline-containing quadruple regimens
  Arms: tinidazole-tetracycline-containing quadruple group

SUMMARY:
The purpose of this study is to assess and compare the effectiveness of levofloxacin-tetracycline -containing and tinidazole-tetracycline-containing quadruple regimens for the primary treatment of Helicobacter pylori infection in patients allergic to penicillin.

DETAILED DESCRIPTION:
Helicobacter pylori(H.pylori), which infects about 50% of the global population, has been recognized as a main risk factor of multiple gastric pathologies, especially non-cardiac gastric cancer. Strongly evidence supports that H.pylori eradication is an effective approach to reduce the incidence of those pathologies.However,Helicobacter pylori eradication is a challenge in patients allergic to penicillin.

Therefore, the investigators aim to assess and compare the effectiveness of levofloxacin-tetracycline -containing and tinidazole-tetracycline-containing quadruple regimens for the primary treatment of Helicobacter pylori infection in patients allergic to penicillin.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 with H. pylori infection.
* Patients Allergic to Penicillin.

Exclusion Criteria:

* Patients with previous H. pylori eradication therapy.
* Patients treated with Histamine-receptor antagonist, proton pump inhibitor, bismuth and antibiotics in the previous 4 weeks.
* Patients with gastrectomy, acute gastrointestinal bleeding and advanced gastric cancer.
* Patients with known or suspected allergy to study medications.
* Currently pregnant or lactating.
* Inability to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Eradication rates in 2 groups | 24 months
  Both intention to treat(ITT) and per-protocol(PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infections in two groups. The ITT analysis includes all randomly assigned patients who take at least one dose of the study medications. The PP analysis is limited to patients who take over 90% of the study medications and complete follow-up.

SECONDARY OUTCOMES:
The rate of improving dyspepsia symptoms after Helicobacter pylori eradication | 24 months
  Dyspepsia symptoms will be measured using a 8-point Likert scale, and patients rate their symptoms from 0 (none) to 8 (severe) before and after the Helicobacter pylori eradication.
The rate of adverse events happening | 24 months
  Similarly, adverse events will also be measured by the Likert scale.
The rate of good compliance | 24 months
  Patients taken over 90% of drugs are considered to have a good compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, PhD,MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu hospital, Jinan, Shandong, China